CLINICAL TRIAL: NCT01610557
Title: A Phase II Randomized Study to Compare Anti-VEGF Agents in the Treatment of Diabetic Macular Edema (CADME)
Brief Title: Ranibizumab and Bevacizumab for Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 120134; 12-EI-0134
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Ranibizumab; Bevacizumab
MeSH Terms: interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series (Experimental): Group 1 eyes were assigned to Ranibizumab-Ranibizumab-Bevacizumab (RRB) treatment sequence and received intravitreal injections of ranibizumab at baseline, Weeks 4, and 8 (period 1), and Weeks 12, 16 and 20 (period 2), then crossed over to receive intravitreal injections of bevacizumab at Weeks 24, 28 and 32 (period 3).
  Participants for whom one eye was enrolled in the study had this eye randomly assigned to one of four groups. Participants for whom both eyes were enrolled had the right eye randomly assigned; the left eye was assigned to the group with the schedule inverse to that for the right eye.
  Interventions: Drug: Ranibizumab; Drug: Bevacizumab
- Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series (Experimental): Group 2 eyes were assigned to Ranibizumab-Bevacizumab-Bevacizumab (RBB) treatment sequence and received intravitreal injections of ranibizumab at baseline and Weeks 4 and 8 (period 1), then crossed over to receive intravitreal injections of bevacizumab at Weeks 12, 16, 20, 24, 28 and 32 (periods 2 and 3).
  Participants for whom one eye was enrolled in the study had this eye randomly assigned to one of four groups. Participants for whom both eyes were enrolled had the right eye randomly assigned; the left eye was assigned to the group with the schedule inverse to that for the right eye.
  Interventions: Drug: Ranibizumab; Drug: Bevacizumab
- Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series (Experimental): Group 3 eyes were assigned to Bevacizumab-Bevacizumab-Ranibizumab (BBR) treatment sequence and received intravitreal injections of bevacizumab at baseline and Weeks 4, 8, 12, 16 and 20 (periods 1 and 2), then crossed over to receive intravitreal injections of ranibizumab at Weeks 24, 28 and 32 (period 3).
  Participants for whom one eye was enrolled in the study had this eye randomly assigned to one of four groups. Participants for whom both eyes were enrolled had the right eye randomly assigned; the left eye was assigned to the group with the schedule inverse to that for the right eye.
  Interventions: Drug: Ranibizumab; Drug: Bevacizumab
- Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series (Experimental): Group 4 eyes were assigned to Bevacizumab-Ranibizumab-Ranibizumab (BRR) treatment sequence and received intravitreal injections of bevacizumab at baseline and Weeks 4 and 8 (period 1), then crossed over to receive intravitreal injections of ranibizumab at Weeks 12, 16, 20, 24, 28 and 32 (periods 2 and 3).
  Participants for whom one eye was enrolled in the study had this eye randomly assigned to one of four groups. Participants for whom both eyes were enrolled had the right eye randomly assigned; the left eye was assigned to the group with the schedule inverse to that for the right eye.
  Interventions: Drug: Ranibizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ranibizumab — Series of three intravitreous injections of ranibizumab (0.3 mg)* or bevacizumab (1.25 mg) administered every 4 weeks for three 12-week periods. Following this crossover phase, eyes received ranibizumab or bevacizumab to which they were originally assigned and treated on an as-needed basis until study completion.
  *Eleven doses of ranibizumab 0.5 mg were given to participants at the start of the study; after FDA approval of the 0.3 mg dose for DME, the protocol was amended and 0.3 mg was used for the remainder of the study (98% of all injections).
Drug: Bevacizumab — Series of three intravitreous injections of ranibizumab (0.3 mg)* or bevacizumab (1.25 mg) administered every 4 weeks for three 12-week periods. Following this crossover phase, eyes received ranibizumab or bevacizumab to which they were originally assigned and treated on an as-needed basis until study completion.
  *Eleven doses of ranibizumab 0.5 mg were given to participants at the start of the study; after FDA approval of the 0.3 mg dose for DME, the protocol was amended and 0.3 mg was used for the remainder of the study (98% of all injections).

SUMMARY:
Background:

* Diabetic macular edema is a common eye complication of diabetes. It causes the blood vessels in the retina at the back of the eye to leak, causing swelling. The macula is the center part of the retina that is important for seeing fine details and for tasks such as reading, driving, or sewing. Swelling of the macula leads to vision loss and possible blindness. Inflammation may play a role in diabetic macular edema. It is also possible that there is a problem with the blood vessels and the blood supply to cells of the retina.
* A chemical in the body called vascular endothelial growth factor (VEGF) is important in the formation of blood vessels in the body. Lowering VEGF levels may help treat diabetic macular edema by reducing abnormal leaking blood vessels in the eye. Drugs that can lower or block VEGF include ranibizumab and bevacizumab. Both drugs have been shown to help treat diabetic macular edema. Researchers want to see if one of the drugs works better than the other.

Objective: To compare the effectiveness of ranibizumab and bevacizumab injections for diabetic macular edema.

Eligibility: Individuals at least 18 years of age who have diabetic macular edema in at least one eye.

Design:

* Participants will be screened with a physical exam and medical history. A full eye exam will be performed. Blood and urine samples will be collected.
* One eye will be selected as the study eye to receive treatment. If both eyes are affected, both eyes may be enrolled in the study and receive different drug treatments.
* The main part of the study will last for 9 months. At each study visit, participants will have physical exams and eye exams. They will answer questions about their health and any side effects from the drugs.
* Participants will be assigned to one of four groups. Two groups will have two series of ranibizumab and one series of bevacizumab shots. The other two groups will have two series of bevacizumab and one series of ranibizumab shots. A series is three eye injections of the same drug every 4 weeks. The injections will be given at these study visits. The series order will vary for the different groups.
* After 9 months, participants will continue to have additional study visits. If the treatment seems to be successful, the study doctor may increase the time between visits. Study injections may be given as needed every 4 weeks for up to 3 years.
* Participants may have laser treatments in a study eye if needed. After being in the study for 1 year, they may also have steroid injections or other treatments as directed for the macular edema.

DETAILED DESCRIPTION:
Objective: Diabetic retinopathy (DR) remains a leading cause of visual impairment. A frequent manifestation of DR is diabetic macular edema (DME) for which laser photocoagulation has been the only proven treatment for the last several decades. Studies have shown that anti-vascular endothelial growth factor (VEGF) injections such as bevacizumab or ranibizumab have been efficacious in treating patients with DME. However, there has been no direct comparison of these agents to determine whether one treatment is more effective than the other. The objective of this study is to compare the treatment efficacy of ranibizumab versus bevacizumab in eyes with DME.

Study Population: Sixty (60) participants with macular edema secondary to diabetes and any stage of DR (other than those requiring scatter laser photocoagulation for proliferative DR) in one or both eyes will be enrolled in this randomized study.

Design: In this Phase II, multi-center, comparative, double-masked study, eyes will be randomly assigned to receive ranibizumab or bevacizumab. During the initial phase of the study participants will participate in a three-period, 36-week, crossover study in which study eyes will be assigned to one of four treatment groups (i.e., treatment sequences). The two drugs and three periods form a RRB/RBB/BBR/BRR pattern as follows:

* Group 1 (RRB pattern) eyes will receive a series of intravitreal injections of ranibizumab at baseline and Weeks 4, 8, 12, 16 and 20, then crossover to receive a series of intravitreal injections of bevacizumab at Weeks 24, 28 and 32.
* Group 2 (RBB pattern) eyes will receive a series of intravitreal injections of ranibizumab at baseline and Weeks 4 and 8, then crossover to receive a series of intravitreal injections of bevacizumab at Weeks 12, 16, 20, 24, 28 and 32.
* Group 3 (BBR pattern) eyes will receive a series of intravitreal injections of bevacizumab at baseline and Weeks 4, 8, 12, 16 and 20, then crossover to receive a series of intravitreal injections of ranibizumab at Weeks 24, 28 and 32.
* Group 4 (BRR pattern) eyes will receive a series of intravitreal injections of bevacizumab at baseline and Weeks 4 and 8, then crossover to receive a series of intravitreal injections of ranibizumab at Weeks 12, 16, 20, 24, 28 and 32.

Participants for whom one eye is enrolled in the study will have this eye randomly assigned to one of the four groups above. Participants for whom both eyes are enrolled in the study will have the right eye randomly assigned to one of the four groups above; the left eye will be assigned to the group with the schedule inverse to that for the right eye. For example, if the right eye is randomly assigned to Group 1 (RRB pattern), the left eye will be automatically assigned to Group 3 (BBR pattern). Thus, at each treatment, the right eye for a participant enrolling both eyes in the study will always receive a different investigational product than the left eye. Following this crossover phase, eyes will be returned to the treatment (ranibizumab or bevacizumab) to which they were originally assigned and treated on an as-needed basis through a common termination date one year from enrollment of the last-enrolled participant at the National Eye Institute (NEI) and through Year 1 at the Bristol Eye Hospital (BEH). Both the treating investigators and participants will be masked to the group assignments. The primary outcome will be assessed at Weeks 12, 24, 36 and Year 1.

Outcome Measures: The primary outcome measure is the mean change in Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity (BCVA). Changes in BCVA from baseline to four weeks following the end of each of the three periods (i.e., Weeks 12, 24 and 36) and at Year 1 will be used for the primary analysis.

Secondary outcomes (assessed between the baseline and Week 12 visits, Weeks 12 and 24 visits and Weeks 24 and 36 visits and at Year 1) will include the mean changes in central macular thickness and central retinal volume by treatment group as measured by optical coherence tomography (OCT); the slope of the changes in BCVA, central macular thickness and retinal volume; the proportion of eyes with visual improvement ≥ 10 letters; the proportion of eyes with visual improvement ≥ 15 letters; the proportion of eyes with ≥ 0.1 log unit loss or gain in logOCT; the proportion of eyes with ≥ 0.05 log unit loss or gain in logOCT; changes in fluid leakage in the macula as demonstrated by fluorescein angiography; and changes in macular structural improvement (i.e., resolution of cystic changes) as measured by OCT. The digital OCT images collected between the Baseline and Week 36 visits will be graded by a masked, external Reading Center.

Other secondary outcomes will include the proportion of eyes meeting criteria for significant worsening, treatment success, or treatment failure, the frequency of re-injection among eyes in the treatment-as-needed phase of the study, and the proportion of eyes receiving focal/grid laser photocoagulation or other adjuvant treatment during the course of the study.

Safety outcomes include the number and severity of adverse events. The number of eyes withdrawn from the investigational product due to vision loss or adverse events and the number of eyes deemed to have worsening disease will also contribute to the assessment of safety.

ELIGIBILITY:
INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant is 18 years of age or older.
2. Participant has a diagnosis of diabetic mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes;
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes;
   * Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria.
3. Participant must understand and sign the protocol's informed consent document.
4. Female participants of childbearing potential must not be pregnant or breast-feeding and must have a negative pregnancy test at screening and must agree to pregnancy testing throughout the study.
5. Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for four weeks after their last injection. Acceptable methods of contraception include:

   * Hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
   * Intrauterine device,
   * Barrier methods (i.e., diaphragm, condom) with spermicide, or
   * Tubal ligation.
6. Participant has at least one eye that meets the study eye eligibility criteria.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Participant is in another investigational study and actively receiving investigational product for DME.
2. Participant has a known hypersensitivity to sodium fluorescein dye.
3. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
4. Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
5. Participant has a history of liver failure.
6. Participant has a known hypersensitivity to bevacizumab, ranibizumab or any of their components.
7. Participant has a blood pressure of > 180/110 (systolic above 180 OR diastolic above 110).

   --If blood pressure is brought below 180/110 by anti-hypertensive treatment, a patient can become eligible.
8. Participant has a history of treatment with oral steroids (greater than or equal to 10 mg of prednisone daily or equivalent) within three months prior to enrollment. Non-ocular depot and inhaled steroid treatments will not exclude a participant.
9. Participant has a history of treatment with systemic anti-VEGF agents within four weeks prior to enrollment.

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below. Participants for whom both eyes meet all of the inclusion criteria and none of the exclusion criteria listed below may have both eyes enrolled in the study if they and the investigator so choose. If both eyes meet all of the inclusion criteria and none of the exclusion criteria listed below, and if the participant and the investigator decide that only one eye should be enrolled in the study, the study eye will be selected by the investigator in consultation with the participant.

STUDY EYE INCLUSION CRITERIA:

1. Eye has a BCVA ETDRS score between 20/32 and 20/400.
2. Eye has definite retinal thickening or cystic changes due to DME based on clinical exam involving the center of the macula that is not refractory to further therapy as based on the investigator's clinical judgment.
3. Eye has retinal thickness in the central subfield on baseline OCT measurement greater than or equal to 330 microns, as measured by Cirrus OCT.
4. Eye has clear ocular media and adequate pupillary dilation sufficient for adequate fundus photographs.

STUDY EYE EXCLUSION CRITERIA:

1. Eye has macular edema considered to be due to a cause other than diabetes.

   An eye is not eligible if:
   * The macular edema is considered to be related to cataract extraction; or
   * Clinical examination and/or OCT suggest that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema.
2. Eye has an ocular condition present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, non-retinal condition).
3. Eye has an ocular condition present (other than DR) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
4. Eye has a history of panretinal scatter photocoagulation (PRP) within three months prior to enrollment.
5. Eye has a history of prior pars plana vitrectomy prior to enrollment.
6. Eye has a history of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within three months prior to enrollment.
7. Eye has a history of Yttrium-Aluminum-Garnet (YAG) capsulotomy performed within two months prior to enrollment.
8. Eye had laser photocoagulation treatment, or received intravitreal or periocular steroids within three months prior to enrollment.
9. Eye has a history of intravitreal anti-VEGF agents within eight weeks prior to enrollment.
10. Eye has had greater than four intravitreal anti-VEGF injections within one year prior to enrollment.
11. Eye has high-risk proliferative DR requiring laser photocoagulation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Wiley, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Bristol Eye Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Klein R, Knudtson MD, Lee KE, Gangnon R, Klein BE. The Wisconsin Epidemiologic Study of Diabetic Retinopathy XXIII: the twenty-five-year incidence of macular edema in persons with type 1 diabetes. Ophthalmology. 2009 Mar;116(3):497-503. doi: 10.1016/j.ophtha.2008.10.016. Epub 2009 Jan 22. PMID 19167079
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Result] Wiley HE, Thompson DJ, Bailey C, Chew EY, Cukras CA, Jaffe GJ, Lee RW, Loken EK, Meyerle CB, Wong W, Ferris FL 3rd. A Crossover Design for Comparative Efficacy: A 36-Week Randomized Trial of Bevacizumab and Ranibizumab for Diabetic Macular Edema. Ophthalmology. 2016 Apr;123(4):841-9. doi: 10.1016/j.ophtha.2015.11.021. Epub 2016 Feb 10. PMID 26875003
- [Result] Sun JK, Josic K, Melia M, Glassman AR, Bailey C, Chalam KV, Chew EY, Cukras C, Grover S, Jaffe GJ, Lee R, Nielsen JS, Thompson DJS, Wiley HE, Ferris FL 3rd; DRCR Retina Network. Conversion of Central Subfield Thickness Measurements of Diabetic Macular Edema Across Cirrus and Spectralis Optical Coherence Tomography Instruments. Transl Vis Sci Technol. 2021 Dec 1;10(14):34. doi: 10.1167/tvst.10.14.34. PMID 34967834
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-EI-0134.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 participants enrolled: 50 participants had one eye randomly assigned (unilateral participants) and 6 participants had two eyes enrolled (bilateral participants) for a total of 62 eyes analyzed at baseline. Bilateral participants had the right eye randomly assigned; the left eye assigned to the group with the schedule inverse to the right eye.
Groups:
- Ranibizumab/Bevacizumab As Needed: Post-36-Week Extension Phase: Eyes assigned to Group 1 or Group 2 in the crossover phase were injected with ranibizumab on an as-needed basis. Eyes assigned to Group 3 or Group 4 in the crossover phase were injected with bevacizumab on an as-needed basis.
  53 participants attended at least one follow-up visit in the post-36-week extension phase: 49 participants who had one eye enrolled and 4 participants who had two eyes enrolled.
Period: 36-Week Randomized Crossover Phase
Arm/Group | Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series | Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series | Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series | Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series | Ranibizumab/Bevacizumab As Needed
Started | 16 (Participants randomly assigned to Grp 1: 14 unilateral and 2 bilateral (left eye assigned to Grp 3)) | 13 (Participants randomly assigned to Grp 2: 12 unilateral and 1 bilateral (left eye assigned to Grp 4)) | 14 (Participants randomly assigned to Grp 3: 13 unilateral and 1 bilateral (left eye assigned to Grp 1)) | 13 (Participants randomly assigned to Grp 4: 11 unilateral and 2 bilateral (left eye assigned to Grp 2)) | 0 (Not applicable for 36-week double-masked randomized crossover phase)
Completed | 16 | 12 (Unilateral participant unable to return for visits after Wk 4 due to recovery from an adverse event) | 14 | 13 | 0 (Not applicable for 36-week double-masked randomized crossover phase)
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Post-36-Week Extension Phase
Arm/Group | Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series | Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series | Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series | Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series | Ranibizumab/Bevacizumab As Needed
Started | 0 (Not applicable for the post-36-week extension phase) | 0 (Not applicable for the post-36-week extension phase) | 0 (Not applicable for the post-36-week extension phase) | 0 (Not applicable for the post-36-week extension phase) | 55
Completed | 0 (Not applicable for the post-36-week extension phase) | 0 (Not applicable for the post-36-week extension phase) | 0 (Not applicable for the post-36-week extension phase) | 0 (Not applicable for the post-36-week extension phase) | 52 (2 bilateral participants withdrew before their first post-36-week extension visit)
Not Completed | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly.
  Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series | Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series | Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series | Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series | Total
Number analyzed (Participants) | 17 | 15 | 16 | 14 | 62
Age, Continuous [Mean (Full Range); unit: years] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
  years | 62.4 [39 to 85] | 65.9 [39 to 87] | 62.3 [39 to 83] | 61.8 [51 to 82] | 63 [39 to 87]
Sex/Gender, Customized [Number; unit: eyes] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
  eyes
    Female | 4 | 8 | 7 | 5 | 24
    Male | 13 | 7 | 9 | 9 | 38
Race/Ethnicity, Customized [Number; unit: eyes] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
  eyes
    Hispanic or Latino | 2 | 0 | 1 | 0 | 3
    Not Hispanic or Latino | 15 | 15 | 14 | 14 | 58
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: eyes] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes
  eyes
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 1 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 2 | 2 | 2 | 8
    White | 12 | 13 | 11 | 10 | 46
    More than one race | 1 | 0 | 2 | 0 | 3
    Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Diabetes Type [Number; unit: eyes] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes
  eyes
    Diabetes Type 1 | 2 | 2 | 1 | 2 | 7
    Diabetes Type 2 | 15 | 13 | 15 | 12 | 55
Hemoglobin A1C (%) [Mean (Full Range); unit: percentage of glycosylated hemoglobin] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
  percentage of glycosylated hemoglobin | 8.1 [6.2 to 11.5] | 8.4 [5.8 to 12.2] | 7.9 [6.2 to 10.6] | 7.8 [5.8 to 10.3] | 8.1 [5.8 to 12.2]
Best-corrected visual acuity [Mean (Full Range); unit: ETDRS letters] — Best-corrected visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS chart.
  Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
  ETDRS letters | 65 [38 to 78] | 61 [32 to 73] | 65 [44 to 75] | 65 [50 to 78] | 64 [32 to 78]
Optical Coherence Tomography (OCT) Central Subfield Mean Thickness [Mean (Full Range); unit: micrometers] — Participants with both eyes enrolled are counted twice (by eye), once for each of the treatment sequences to which an eye was assigned randomly. Although 56 participants enrolled, 6 participants had two eyes enrolled for a total of 62 eyes.
  Optical Coherence Tomography (OCT) scans were masked and graded at an external reading center (Duke University, Durham, North Carolina).
  micrometers | 484 [334 to 720] | 444 [366 to 602] | 471 [362 to 606] | 508 [358 to 653] | 477 [334 to 720]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) From Baseline to 36 Weeks (Crossover Phase of the Study)
Description: The primary outcome for 3-months change in BCVA utilized data from Weeks 12, 24 and 36 aggregated in a linear mixed-effects model. This model included adjustments accounting for period (i.e., Weeks 12, 24 and 36), treatment in current period, treatment in prior period, and baseline BCVA to provide the estimated 3-month BCVA change.
  Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 36 Weeks
Population: A total of 56 participants (62 eyes) were enrolled and 55 participants (61 eyes) completed the 36-week crossover phase of the study.
Measure: Mean (95% Confidence Interval); unit: ETDRS letters
Units Other Than Participants: eyes
Groups:
- Bevacizumab: Represents the estimated effect of bevacizumab for a 3-month period, adjusted for period and baseline value.
- Ranibizumab: Represents the estimated effect of ranibizumab for a 3-month period, adjusted for period and baseline value.
Arm/Group | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 55 | 55
Number analyzed (eyes) | 61 | 61
ETDRS letters | 5.3 [3.2 to 7.4] | 6.6 [4.5 to 8.7]
Statistical Analysis 1: Comparison: Bevacizumab vs Ranibizumab; Test type: Superiority or Other; p = 0.039, Linear mixed-effects model; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.07 to 2.5] — The difference represents the estimated difference between ranibizumab and bevacizumab, adjusted for baseline visual acuity, study period, and clinical site and a subject effect for eyes nested within subject

2. Secondary Outcome: Change in Central Retinal Thickness Assessed by Optical Coherence Tomography (OCT) Central Subfield Mean Thickness (CSMT) From Baseline to 36 Weeks (Crossover Phase of the Study)
Description: Optical Coherence Tomography (OCT) scans were graded in masked fashion by Duke University Reading Center (Durham, North Carolina). Per the initial protocol specifications, OCT scans were to be performed on a Cirrus OCT machine; however, some scans were performed on a Spectralis OCT machine at one of the sites due to technical difficulties. The protocol was amended to allow for Cirrus and Spectralis OCT scans at subsequent visits at the affected site. Spectralis values were then converted to Cirrus central subfield mean thickness (CSMT) values through a validated linear conversion function.
Time Frame: Baseline and 36 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: micrometers
Units Other Than Participants: eyes
Arm/Group | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 55 | 55
Number analyzed (eyes) | 61 | 61
micrometers | -89 [-116 to -62] | -137 [-164 to -110]
Statistical Analysis 1: Comparison: Bevacizumab vs Ranibizumab; Test type: Superiority or Other; p < 0.001, Linear mixed-effects model; Mean Difference (Final Values) = -48, 95% CI 2-sided [-65 to -31] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Data were collected from 56 participants randomly-assigned to Groups 1 through 4 during the 36-week crossover period. After 36 weeks, data were collected from 53 participants who completed at least one post-36-week visit.
Description: 36-week crossover period:Of the 56 participants, 50 had one eye and 6 had two eyes enrolled; data collected from the 6 participants with two eyes enrolled are reflected in the group to which the participant's right eye was randomly assigned. Post-36-weeks:Of the 53 participants, data were collected from 49 with one eye and 4 with two eyes enrolled.
Groups:
- Ranibizumab As Needed (Post-36-Week Extension): Post-36-Week Extension Phase: Eyes assigned to Group 1 or Group 2 in the crossover phase were injected with ranibizumab on an as-needed basis.
  Participants with one eye assigned in either Group 1 or Group 2 who had at least one follow-up visit in the post-36-week extension are included in the number of participants at risk.
  Participants for whom two eyes were assigned (bilateral participants) are not included.
- Bevacizumab As Needed (Post-36-Week Extension): Post-36-Week Extension Phase: Eyes assigned to Group 3 or Group 4 in the crossover phase were injected with bevacizumab on an as-needed basis.
  Participants with one eye assigned in either Group 3 or Group 4 who had at least one follow-up visit in the post-36-week extension are included in the number of participants at risk.
  Participants for whom two eyes were assigned (bilateral participants) are not included.
- Ranibizumab and Bevacizumab As Needed (Post-36-Week Extension): Post-36-Week Extension Phase: Eyes assigned to Group 1 or Group 2 in the crossover phase were injected with ranibizumab on an as-needed basis. Eyes assigned to Group 3 or Group 4 in the crossover phase were injected with bevacizumab on an as-needed basis.
  Participants with two eyes assigned who had at least one follow-up visit in the post-36-week extension are included in the number of participants at risk.
  Participants for whom one eye was assigned (unilateral participants) are not included.
Arm/Group | Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series | Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series | Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series | Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series | Ranibizumab As Needed (Post-36-Week Extension) | Bevacizumab As Needed (Post-36-Week Extension) | Ranibizumab and Bevacizumab As Needed (Post-36-Week Extension)
Serious Adverse Events (participants affected / at risk) | 3/16 | 1/13 | 1/14 | 1/13 | 1/25 | 0/24 | 0/4
Other Adverse Events (participants affected / at risk) | 13/16 | 12/13 | 9/14 | 9/13 | 13/25 | 12/24 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series (N=16) | Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series (N=13) | Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series (N=14) | Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series (N=13) | Ranibizumab As Needed (Post-36-Week Extension) (N=25) | Bevacizumab As Needed (Post-36-Week Extension) (N=24) | Ranibizumab and Bevacizumab As Needed (Post-36-Week Extension) (N=4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Ranibizumab-Ranibizumab-Bevacizumab Injection Series (N=16) | Group 2 - Ranibizumab-Bevacizumab-Bevacizumab Injection Series (N=13) | Group 3 - Bevacizumab-Bevacizumab-Ranibizumab Injection Series (N=14) | Group 4 - Bevacizumab-Ranibizumab-Ranibizumab Injection Series (N=13) | Ranibizumab As Needed (Post-36-Week Extension) (N=25) | Bevacizumab As Needed (Post-36-Week Extension) (N=24) | Ranibizumab and Bevacizumab As Needed (Post-36-Week Extension) (N=4)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Albumin urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyst removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No outcome data should be presented until after a manuscript is accepted for publication.